CLINICAL TRIAL: NCT01770652
Title: An Open-label Study to Compare the Pharmacokinetic Profiles of a Single Dose of Ferriprox in Subjects With Impaired Renal Function and Healthy Volunteers
Brief Title: An Open-label, Non-randomized, Parallel Group Study in Subjects With Mild, Moderate, Severe, or No Renal Impairment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ApoPharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: LA39-0412
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Renal Impairment
Keywords: Renal Impairment; Kidney Impairment; Kidney Disease; Ferriprox; Deferiprone; DFP (deferiprone); L1
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases | interventions — Deferiprone; Long Interspersed Nucleotide Elements; Isoflurophate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal renal function (Experimental): Healthy volunteers, defined as having an estimated glomerular filtration rate (eGFR) ≥90 mL/min/1.73m^2. All subjects received a single 33 mg/kg oral dose of deferiprone.
  Interventions: Drug: Deferiprone
- Mild Renal Impairment (Experimental): Mild impairment, defined as having an eGFR 60-89 mL/min/1.73m^2. All subjects received a single 33 mg/kg oral dose of deferiprone.
  Interventions: Drug: Deferiprone
- Moderate Renal Impairment (Experimental): Mild impairment, defined as having an eGFR 30-59 mL/min/1.73m^2. All subjects received a single 33 mg/kg oral dose of deferiprone.
  Interventions: Drug: Deferiprone
- Severe Renal Impairment (Experimental): Severe impairment, defined as having an eGFR 15-19 mL/min/1.73m^2. All subjects received a single 33 mg/kg oral dose of deferiprone.
  Interventions: Drug: Deferiprone

INTERVENTIONS:
Drug: Deferiprone — Oral iron chelator
  Other Names: Ferriprox; L1; DFP

SUMMARY:
Multi-center, non-randomized, open-label, single-dose, parallel group study to determine the effect of impaired renal function on the PK of deferiprone and its 3-O-glucuronide metabolite following a single oral dose of 33mg/kg Ferriprox®.

DETAILED DESCRIPTION:
Post-marketing study to evaluate the effect of impaired renal function on the pharmacokinetics (PK) of deferiprone and its 3-O-glucuronide metabolite and on the safety of Ferriprox® in subjects with mild, moderate and severe renal impairment as compared to healthy volunteers.

ELIGIBILITY:
Main Inclusion Criteria:

All subjects:

1. Adult males or females, 18 - 75 years of age (inclusive);
2. Body weight ≥ 45 kg;
3. Body mass index (BMI) range of approximately 18.5-32 kg/m^2 (inclusive);
4. Absolute neutrophil count (ANC) of >1.5x10^9/L;

Healthy volunteers:

1. Medically healthy with clinically insignificant screening results (e.g., laboratory profiles, medical history, vital signs, physical examination);
2. eGFR ≥ 90 mL/min/1.73m^2;

Renally impaired subjects:

1. Considered clinically stable in the opinion of the Investigator;
2. Subjects with mild renal impairment (eGFR 60-89 mL/min/1.73m^E2) OR moderate renal impairment (eGFR 30-59 mL/min/1.73m^2) OR severe renal impairment (eGFR 15-29 mL/min/1.73m^2).

Main Exclusion Criteria:

1. History of renal transplant;
2. Subjects undergoing any method of dialysis;
3. History or presence of clinically unstable significant respiratory, cardiovascular, pulmonary, hepatic, renal (except for subjects assigned to one of the renally impaired groups), hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease;
4. Disorders or surgery of the gastrointestinal tract which may interfere with drug absorption or may otherwise influence the PK of the investigational medicinal product (e.g. cholecystectomy, resections of the small or large intestine, febrile conditions, chronic diarrhea, chronic vomiting, endocrine disease, severe infections, acute inflammations, etc.);
5. Clinically significant abnormalities on 12-lead ECG (e.g., QTcF≥430 ms in males or ≥450 ms in females);
6. Evidence of liver damage: hepatitis B and C; aspartate aminotransferase (AST), alanine aminotransferase (ALT) that is considered clinically significant by the Investigator;
7. Participation in another clinical trial within 28 days prior to the study drug administration;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Tricta, MD, Study Chair — ApoPharma
Locations (2):
- Canada (2):
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Algorithme Pharma Inc., Mount Royal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Hepatic Function (Healthy Volunteers): Healthy volunteers as defined by an eGFR ≥90 mL/min/1.73m^2 as determined by the estimated glomerular filtration rate (eGFR) from the Modification of Diet in Renal Disease (MDRD) Study will receive a single 33mg/kg oral dose of deferiprone.
  Deferiprone
- Mild Renal Impairment: Mild renal impairment defined as eGFR 60-89 mL/min/1.73m^2 as determined by the estimated glomerular filtration rate (eGFR) from the Modification of Diet in Renal Disease (MDRD) Study will receive a single 33mg/kg oral dose of deferiprone.
  Deferiprone
- Moderate Renal Impairment: Moderate renal impairment as defined by eGFR 30-59 mL/min/1.73m^2 as determined by the estimated glomerular filtration rate (eGFR) from the Modification of Diet in Renal Disease (MDRD) Study will receive a single 33mg/kg oral dose of deferiprone.
  Deferiprone
- Severe Renal Impairment: Severe renal impairment as defined by an eGFR 15-19 mL/min/1.73m^2 as determined by the estimated glomerular filtration rate (eGFR) from the Modification of Diet in Renal Disease (MDRD) Study will receive a single 33mg/kg oral dose of deferiprone.
  Deferiprone
Period: Overall Study
Arm/Group | Normal Hepatic Function (Healthy Volunteers) | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Hepatic Function (Healthy Volunteers) | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 4 | 6 | 23
  >=65 years | 1 | 2 | 4 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 3 | 2 | 13
  Male | 3 | 5 | 5 | 6 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 0 | 2
  White | 8 | 6 | 8 | 8 | 30
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 8 | 8 | 8 | 32
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 8 | 8 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cmax for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: Cmax was assessed over a 24-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite in subjects with normal, mild, moderate and severe renal impairment. Blood samples were obtained prior to dosing and at 0.25, 0.50, 0.75, 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 9, 12, 16, and 24 hours post-dose.
Time Frame: 24-hour interval
Population: The pharmacokinetic population included all subjects who had sufficient data to derive the value of at least one pharmacokinetic parameter.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Normal Renal Function (Healthy Volunteers): Healthy volunteers as defined by an eGFR ≥90 mL/min/1.73m^2 as determined by the estimated glomerular filtration rate (eGFR) from the Modification of Diet in Renal Disease (MDRD) Study will receive a single 33mg/kg oral dose of deferiprone.
  Deferiprone
Arm/Group | Normal Renal Function (Healthy Volunteers) | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
μg/mL
  Cmax for serum deferiprone | 37.1 (12.0) | 33.4 (9.5) | 43.3 (22.9) | 30.6 (16.2)
  Cmax for serum deferiprone-3-o-glucuronide | 47.8 (6.2) | 60.8 (10.3) | 118.8 (48.3) | 150.8 (32.4)

2. Secondary Outcome: Safety and Tolerability of Ferriprox® in Subjects With Renal Impairment.
Description: The number of participants who experienced adverse events (including any changes of clinical significance in physical examinations, vital signs, 12-lead ECG, and clinical laboratory tests) following a single dose of Ferriprox.
Time Frame: From time of dosing until 72 hours post-dose
Measure: Number; unit: participants
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
participants | 2 | 5 | 1 | 1

3. Primary Outcome: Tmax for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: Tmax was assessed over a 24-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite. Blood samples were obtained prior to dosing and at 0.25, 0.50, 0.75, 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 9, 12, 16, and 24 hours post-dose.
  The results of the Tmax parameter are reported as the median and range (other parameters are reported as mean and standard deviation).
Time Frame: 24 hour interval
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour
  Tmax for Serum Deferiprone | 0.50 [0.25 to 1.00] | 0.75 [0.50 to 1.00] | 1.00 [0.50 to 2.00] | 0.75 [0.25 to 4.00]
  Tmax for Serum Deferiprone 3-O-glucuronide | 2.50 [1.33 to 3.00] | 2.50 [2.00 to 3.00] | 3.00 [2.00 to 6.00] | 4.00 [2.00 to 6.00]

4. Primary Outcome: AUC Zero to Infinity (AUC0-∞) for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: AUC0-∞ was assessed over a 24-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite. Blood samples were obtained prior to dosing and at 0.25, 0.50, 0.75, 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 9, 12, 16, and 24 hours post-dose.
Time Frame: 24 hour interval
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
μg*h/mL
  AUC0-∞ for serum deferiprone 3-O-Glucuronide | 78.1 (27.8) | 76.9 (15.7) | 74.9 (15.1) | 70.9 (8.5)
  AUC0-∞ for serum deferiprone | 252.6 (35.4) | 319.1 (54.1) | 703.2 (229.6) | 1438.5 (335.5)

5. Primary Outcome: T1/2 for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: T1/2 was assessed over a 24-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite. Blood samples were obtained prior to dosing and at 0.25, 0.50, 0.75, 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 9, 12, 16, and 24 hours post-dose.
Time Frame: 24 hour interval
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
hour
  T1/2 for Serum Deferiprone | 1.68 (0.27) | 1.77 (0.17) | 2.03 (0.32) | 2.20 (0.91)
  T1/2 for Serum Deferiprone 3-O-Glucuronide | 2.14 (0.32) | 2.58 (0.45) | 2.58 (0.38) | 3.35 (0.48)

6. Primary Outcome: Ae24 for Urine Deferiprone and Deferiprone 3-O-glucuronide
Description: Ae24 (the amount excreted in urine from time zero to 24 hours) was assessed over a 24-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite. Urine samples were collected at the intervals of -2 to 0 hours pre-dose and 0 to 2, 2 to 4, 4 to 8, 8 to 12, and 12 to 24 hours post-dose.
Time Frame: 24 hour interval
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
mg
  Ae24 for urine deferiprone | 78 (33) | 69 (20) | 36 (12) | 24 (10)
  e24 for urine deferiprone 3-O-Glucuronide | 5987 (1332) | 6608 (1630) | 5812 (929) | 5318 (1683)

7. Primary Outcome: Fe24 for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: Fe24 (fraction of dose excreted in urine from time zero to 24 hours) was assessed over a 24-hour interval for analyses of deferiprone and its 3-O-glucuronide metabolite. Urine samples were collected at the intervals of -2 to 0 hours pre-dose and 0 to 2, 2 to 4, 4 to 8, 8 to 12, and 12 to 24 hours post-dose.
  Some of the Fe24 values were over 100% which could be explained by variability in urine collection (e.g. incomplete collection of urine into the container) and volume measurement, as well as analytical imprecision.
Time Frame: 24-hour interval
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of dose excreted in urine from 0-24 hr
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 8 | 8 | 8 | 8
% of dose excreted in urine from 0-24 hr
  Fe24 for urine deferiprone | 3.5 (1.6) | 2.9 (0.6) | 1.5 (0.5) | 1.0 (0.4)
  Fe24 for urine deferiprone 3-O-glucuronide | 115.0 (16.2) | 123.2 (12.7) | 104.5 (11.6) | 97.9 (28.5)

ADVERSE EVENTS:
Time Frame: Up to 4 days: from the time of administration of study drug until a follow-up telephone call 48 to 72 hours after discharge
Arm/Group | Normal Hepatic Function (Healthy Volunteers) | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/8 | 5/8 | 1/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Hepatic Function (Healthy Volunteers) (N=8) | Mild Renal Impairment (N=8) | Moderate Renal Impairment (N=8) | Severe Renal Impairment (N=8)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Soft stool
Somnolence (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Cramp in right calf
Dysuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — Difficulty urinating
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Metallic taste in mouth
Chills (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Shivering

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less